CLINICAL TRIAL: NCT01098318
Title: Rhodiola Rosea Therapy of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT005230; R21AT005230 (NIH)
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Depression
Keywords: Depression; Antidepressant Therapy; Herbal Treatment; Rhodiola rosea; Alternative Therapy
MeSH Terms: conditions — Depression | interventions — Sertraline; Refit milk powder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rhodiola rosea (Experimental): Herbal extract
  Interventions: Dietary Supplement: Herbal extract
- Sertraline (Active Comparator): Conventional anti-depressant
  Interventions: Drug: Sertraline
- Sugar pill (Placebo Comparator): Lactose monohydrate
  Interventions: Other: Lactose monohydrate

INTERVENTIONS:
Dietary Supplement: Herbal extract — 340-1,360 mg daily
  Other Names: Golden root
  Arms: Rhodiola rosea
Drug: Sertraline — 50-200 mg daily
  Other Names: Zoloft
  Arms: Sertraline
Other: Lactose monohydrate — 1-4 capsules daily
  Other Names: Milk powder
  Arms: Sugar pill

SUMMARY:
Prior research has shown that Rhodiola rosea may be an effective, short-term, anti-depressant therapy. This study will examine the anti-depressant effect of Rhodiola rosea vs. a conventional, anti-depressant drug in the treatment of major depression.

DETAILED DESCRIPTION:
We will study the antidepressant action of R. rosea in patients with MDD. Depression affects more than a billion people world wide, and is now recognized as one of the most disabling medical conditions. It accounts for more than 11% of the total disease burden worldwide, and can result in devastating consequences and functional impairment exceeded only by that of cancer and cardiovascular disease. It results in substantial social, occupational, and personal disability and in increased medical co-morbidity and death by suicide. It is considered to be a multi-systemic disorder characterized by neurotransmitter, neuroendocrine, immunologic, and autonomic, and infectious disturbances. Although the development of antidepressant drug therapy has simplified the treatment of MDD, a substantial segment of the world's population remains untreated for economic, cultural, or personal reasons. As a result, many individuals seek CAM for relief of their symptoms. The identification of effective CAM therapies for MDD is of public health relevance. R. rosea belongs to the family Crassulaceae, and has a long history as a folk remedy for enhancing physical and emotional endurance. Its adaptogen, or preventive, properties have also led to its use in treating cancer, infection, depression, and other nervous system disorders. Several animal and human studies suggest that R. rosea may have antidepressant properties. For specific aim #1, we will ask: Is R. rosea a safe and effective short-term therapy (vs. sertraline and placebo) for patients with MDD?" To answer this question, patients meeting DSM IV criteria for mild to moderate MDD will be enrolled in a 12-week, randomized, double-blind, placebo-controlled, parallel group, dose-escalation study of R. rosea extract 340-1,360 mg daily vs. sertraline 50-200 mg daily. The primary outcome measure will be change over time in the 17-item Hamilton Depression Rating score. We hypothesize that R. rosea will have superior efficacy vs. placebo and comparable efficacy vs. sertraline. For specific aim #2, we will ask: Does R. rosea therapy result in a favorable tolerability and quality of life (QOL) profile vs. sertraline and placebo? To answer this question, we will obtain safety and QOL measures across treatment conditions that include: (i) frequency, duration, and severity of adverse events, (ii) frequency of serious adverse events, (iii) frequency of dosage reduction, (iv) frequency of treatment discontinuation, and (v) QOL and sexual performance measures. We hypothesize that R. rosea will have a superior tolerability profile vs. sertraline, and similar tolerability vs. placebo. We further hypothesize that R. rosea will have superior QOL and sexual performance ratings vs. sertraline and placebo. Results from this study will be used to inform future research hypotheses and to estimate the effect size necessary to power a future, large scale study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (all races and ethnicity) ≥ 18 years old
* DSM IV Axis I diagnosis of mild to moderate Major Depressive Disorder
* Baseline CGI/S rating of 3 ('mild') or 4 ('moderate')
* Baseline Hamilton Depression Rating score ≥ 10
* Not receiving other antidepressant therapy
* Able to provide signed informed consent

Exclusion Criteria:

* Patients < 18 years old
* Current primary DSM IV Axis I diagnosis other than Major Depressive Disorder
* CGI/S rating of 5 ('marked'), 6 ('severe') or 7 ('very severe')
* Actively suicidal or requiring hospitalization
* Uncontrolled medical condition
* Pregnant or nursing women
* Women of child-bearing potential not using a medically acceptable form of contraception
* Concurrent use of herbal remedies or mineral supplements [Note: Use of mineral supplements prescribed for medical purposes (e.g., osteoporosis) will not be excluded]
* Current use of chemotherapy or other medication (e.g., interferon) known to produce fatigue or mood changes
* Known sensitivity to R. rosea or sertraline
* History of non-response to sertraline in the current depressive episode

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun J. Mao, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mao JJ, Xie SX, Zee J, Soeller I, Li QS, Rockwell K, Amsterdam JD. Rhodiola rosea versus sertraline for major depressive disorder: A randomized placebo-controlled trial. Phytomedicine. 2015 Mar 15;22(3):394-9. doi: 10.1016/j.phymed.2015.01.010. Epub 2015 Feb 23. PMID 25837277
- See also: Depression Research Unit-Department of Psychiatry Clinical Research Programs — http://www.med.upenn.edu/psychiatry/programs.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There are actually 58 subjects who signed consents. However, one subject withdrew consent immediately after signed it due to change of mind. This subject didn't take any medication, therefore, only 57 subject received study intervention.
Period: Overall Study
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Started | 20 | 19 | 18
Completed | 17 | 12 | 15
Not Completed | 3 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill | Total
Number analyzed (Participants) | 20 | 19 | 18 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (16.9) | 41.4 (14.6) | 46.7 (15.2) | 45.0 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 8 | 26
  Male | 12 | 9 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms as Measured by the Hamilton Depression Rating Scale (17-items) at Week 8 and Week 12.
Description: Hamilton Depression Rating Scale (HAM-D) is a validated, clinician-rated instrument for ascertaining the severity of MDD symptoms. The 28-item Hamilton Depression Rating Scale was used to determine the primary outcome of 17-item HAM-D score. The HAM-D will serves as the primary outcome measure. HAM-D17 score ranges from 0 to 68. Higher score indicates more depressed symptom.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Number analyzed (Participants) | 20 | 19 | 18
units on a scale
  HAM-D17@WK8 | 8 (5.4) | 8.3 (4.5) | 8.9 (6.5)
  HAM-D17@WK12 | 7.9 (6) | 7.8 (4.3) | 8.5 (6.7)

2. Secondary Outcome: The Clinical Global Impression (CGI) Severity and Change
Description: A clinician-rated measure of global symptom severity (CGI/S) and symptom change (CGI/C) of MDD. Severity was rated as "Not ill"; "Borderline ill"; "Mild"; "Moderate"; "Moderately severe"; "Severe" and "Extremely severe". Global change was rates as "Very much improved"; "Much improved"; "Minimally improved"; "Unchanged";"Minimally worse";"Much worse" and "Very much worse". Here in severity, we reported the N(%) of subjects who were not ill or borderline ill. In change, we reported N(%) of subjects who were "Very much improved" or "Much imp[roved".Subjects started the study with mild to moderate MDD (moderate or above rating in the CGI-S). At WK12, the #/% of subjects in each treatment group who were not ill at WK12 (CGI-S) and who had much improved or very much improved at WK12 (CGI-C) was reported.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Number analyzed (Participants) | 20 | 19 | 18
Participants
  WK12 CGI-Severity (Not ill and Borderline ill) | 9 | 6 | 7
  WK12 CGI-C (Much improved and very much improved) | 10 | 7 | 7

3. Secondary Outcome: Change in Depressive Symptoms as Measured by the Beck Depression Inventory
Description: All enrolled subjects were analyzed. Mean change in Beck Depression Inventory (BDI) total scores were reported. BDI is a self-reported outcome measuring the severity of depression. A negative # means a reduction in BDI score at the end of treatment compared to baseline which represents an improvement in depression symptoms. BDI total score ranges from 0-63. BDI score of 1-16 represents low level of depression;17-30 represents moderate level of depression; >=31 represents significant level of depression. A reduction in the BDI score represents improvement in the depression symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Number analyzed (Participants) | 20 | 19 | 18
scores on a scale | -14.0 (10.0) | -13.7 (5.1) | -7.5 (12.2)

4. Secondary Outcome: Change in Sexual Function
Description: This is a patient completed rating of sexual function and satisfaction. It is used to assess current sexual health and changes in sexual health over time measured by the overall sexual satisfaction score. The reported score is the overall degree of sexual satisfaction attained. The score ranges from 0 to 100. Higher score indicates more sexual satisfaction.
Time Frame: 12 weeks
Population: All enrolled subjects were analyzed
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Number analyzed (Participants) | 20 | 19 | 18
scores on a scale
  Baseline | 48 [10 to 83] | 36 [5 to 62] | 17 [5 to 31]
  WK12 | 49 [18 to 77] | 25.5 [14 to 37] | 12 [6 to 45]

5. Secondary Outcome: Number of Participants With Suicide Ideation as Determined by the Columbia Suicide Form
Description: Descriptive analysis of number of subjects in each treatment group who had suicidal ideation at baseline and WK12.
Time Frame: 12 weeks
Population: All enrolled subjects were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Number analyzed (Participants) | 20 | 19 | 18
Participants
  Baseline | 6 | 6 | 9
  WK12 | 0 | 0 | 2

6. Secondary Outcome: Number of Participants With Treatment Emergent Side Effects
Time Frame: 12 weeks
Population: All enrolled subjects were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Number analyzed (Participants) | 20 | 19 | 18
Participants | 6 | 12 | 3

ADVERSE EVENTS:
Arm/Group | Rhodiola Rosea | Sertraline | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 6/20 | 12/19 | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rhodiola Rosea (N=20) | Sertraline (N=19) | Sugar Pill (N=18)
Sexual dysfunction (General disorders) | 1 (1) | 4 (7) | 0 (0)
Nervousness (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (10) | 1 (1)
Dizziness (General disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Subjects refuse to answer measures such as the RUSH sexual inventory and the CSSR. Therefore, no statistical analysis was performed on these. In addition, suicidal ideation (measured by CSSR) was captured in the AE form during the study peiod.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No